CLINICAL TRIAL: NCT05729880
Title: Can Ultrasound be Used as a Measure of Muscle Quality? A Validation Study Comparing Ultrasound With MRI and MRS in Older and Younger Persons.
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-22-44
Record Dates: First submitted 2023-01-16; First posted 2023-02-15 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Muscle Atrophy
Keywords: ultrasound; mri
MeSH Terms: conditions — Muscular Atrophy | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older: 16 older (>50y) will be recruited. MRI, MRS and Ultrasound will be measured in each participant in calf and thigh muscle, at the same location within a 1 hour time frame.
  Interventions: Diagnostic Test: MRI, MRS; Diagnostic Test: Ultrasound
- Young: 16 young (<40y) will be recruited. MRI, MRS and Ultrasound will be measured in each participant in calf and thigh muscle, at the same location within a 1 hour time frame.
  Interventions: Diagnostic Test: MRI, MRS; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: MRI, MRS — Scan of right calf and thigh
Diagnostic Test: Ultrasound — Scan of right calf and thigh

SUMMARY:
This study aims to see if ultrasound can be used as a reliable and valid method to measure fatty infiltration, muscle thickness and muscle architecture to provide a quick, cheap and mobile alternative measure of muscle quality to MRI.

The MRS and MRI images will be used to validate the ultrasound images.

DETAILED DESCRIPTION:
A key hallmark of the natural biology of ageing is a progressive loss of skeletal muscle mass, strength and aerobic capacity, termed 'sarcopenia' (Cruz-Jentoft et al. 2019a). The association between muscle loss (mass and quality) and increased incidence of falls, fractures, metabolic disease and other health complications is well established. Despite exercise and physiotherapy, recovery from these is often incomplete and studies have failed to identify fully effective countermeasures (Reeves et al, 2005). Ways to objectively measure the clinical effectiveness of the countermeasures are also limited.

Muscle quality can be measured in terms of muscle thickness, architecture (pennation angle and fascicle length) and fatty infiltration. At present ultrasound muscle thickness and architecture have been shown against MRI to be a reliable and valid but fatty infiltration can only be measured reliably using MRI. MRI is an expensive, time consuming and immobile technique limiting its use as a clinical tool in a rehabilitative setting. Finding a cheaper, quicker and mobile alternative, such as ultrasound, would enable clinicians to gather useful information on patient muscle quality in an objective manner and use this information to tailor treatment accordingly.

15 old (>50y) and 15 young (<40y) will be recruited. MRI, MRS and Ultrasound will be measured in each participant in calf and thigh muscle, at the same location within a 1 hour time frame.

MRI and MRS will provide the validation to ultrasound fatty infiltration.

ELIGIBILITY:
Inclusion Criteria:

- Age <40y or >50yrs

Exclusion Criteria:

1. Significant cognitive deficits and the inability to follow directions during assessment.
2. Neurological, neuromuscular, or musculoskeletal disorders that could impair the quality of the muscle. eg. CP, muscular dystrophy or SCI
3. Prosthesis with metalwork, eg. metal work from surgery
4. Aneurysm clip in situ
5. No metal work anywhere, history of metal fragments in eyes, spinal cord or brain.
6. Previous exposure to metal flakes and metallic injury.
7. No external implants; cochlear implant, spinal cord simulator, pacemaker or other implanted electronic devices.
8. Non-removal hearing aids
9. FEMALE ONLY Not pregnant
10. Not claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound muscle thickness (cm) | 1 year
  A single ultrasound image can measure both thickness (cm) and echogenecity (AU). Echogenecity has been used as a proxy for fat infiltration. By combining both thickness and fat infiltration and index of muscle quality can be determined
Ultrasound echogenecity (arbitrary units on histogram) | 1 year
  A single ultrasound image can measure both thickness (cm) and echogenecity (AU). Echogenecity has been used as a proxy for fat infiltration. By combining both thickness and fat infiltration and index of muscle quality can be determined
Fat fraction | 1 year
  Obtained from MRI and will be used to validate the ultrasound echogenecity

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- University, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared.